CLINICAL TRIAL: NCT00347178
Title: Prophylactic Laser Iridotomy for Eyes With Narrow Drainage Angles; A Randomised Controlled Trial
Brief Title: Asymptomatic Narrow Angles - Laser Iridotomy Study; Multicentric RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Singapore National Eye Centre (Other Government)
Collaborators: National Medical Research Council (NMRC), Singapore (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R358/16/2004
Record Dates: First submitted 2006-06-30; First posted 2006-07-04 (Estimated); Last update posted 2006-07-04 (Estimated); Status verified 2006-06

CONDITIONS: Asymptomatic Narrow Angles; Primary Angle Closure Suspects
Keywords: Asymptomatic Narrow Angles; Primary Angle Closure Suspects; Laser Peripheral Iridotomy; Randomised Controlled Trial

INTERVENTIONS:
Procedure: Laser Peripheral Iridotomy

SUMMARY:
This is a multicentric, randomised, controlled study comparing Laser Iridotomy (LI) to no treatment in subjects with asymptomatic narrow angles (ANA).One eye of each subject with ANA will be randomised to undergo LI and the other eye will be left alone and will serve as an internal control. Subjects are proposed to be followed up once a year for 5 years.

DETAILED DESCRIPTION:
Objective: This study will compare LI versus no treatment in subjects with asymptomatic narrow angles, the anatomical trait that predisposes to primary angle closure glaucoma (PACG), in order to assess the effectiveness of prophylactic treatment in the prevention of blindness due to PACG.

Eligibility: 1. Bilateral Narrow angles; 2. Age 50 years and above; 3. Informed consent obtained prior to or at baseline visit.

Trial Design: Subjects with asymptomatic ANA undergoes randomisation after comprehensive ocular exam followed by randomisation to LI in one eye and no treatment in the other eye. Follow up is done for 5 years with yearly examination.

ELIGIBILITY:
Inclusion Criteria:

1. Bilateral Narrow angles
2. Age 50 years and above
3. Informed consent obtained prior to or at baseline visit

Exclusion Criteria:

1. Presence of PAS
2. IOP > 21 mm Hg
3. Glaucomatous optic neuropathy and/or CDR > 0.7
4. Secondary angle closure such as uveitis, neovascularisation etc.
5. Prior intraocular surgery or penetrating eye injury
6. Corneal disorders such as corneal endothelial dystrophy except mild corneal guttae
7. Evidence of prior acute angle closure event
8. High risk of acute angle closure.
9. Significant cataract and visual acuity less than 20/40
10. Constant use of contact lens for refractive correction
11. Chronic use of topical or systemic steroids
12. Established retinopathies on ocular treatments (e.g. Diabetic)
13. Any other disease which is likely to cause field loss in next 3 years
14. Severe health problems decreasing life expectancy to less than one year.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 544
Dates: Start 2005-01; Study Completion 2013-01

PRIMARY OUTCOMES:
Peripheral anterior synechiae formation
IOP elevation >21 mm Hg
Development of acute angle closure event

SECONDARY OUTCOMES:
Changes in the grading of Modified Schaffer Grading
Development of glaucomatous optic neuropathy
Development of corresponding visual field loss by automated perimetry
Change in HRT optic disc parameters
Change in UBM angle parameters
Formation of disc pallor

CONTACTS AND LOCATIONS:
Overall Officials: Tin - Aung, FRCSEd PhD, Principal Investigator — Singapoe National Eye Centre
Locations (1):
- Singapore Eye Research Institute, Singapore, Singapore

REFERENCES:
- [Derived] Baskaran M, Kumar RS, Friedman DS, Lu QS, Wong HT, Chew PTK, Lavanya R, Narayanaswamy A, Perera SA, Foster PJ, Aung T. The Singapore Asymptomatic Narrow Angles Laser Iridotomy Study: Five-Year Results of a Randomized Controlled Trial. Ophthalmology. 2022 Feb;129(2):147-158. doi: 10.1016/j.ophtha.2021.08.017. Epub 2021 Aug 26. PMID 34453952
- [Derived] Narayanaswamy A, Baskaran M, Tun TA, Htoon HM, Aung T. Effect of Pharmacological Pupil Dilatation on Angle Configuration in Untreated Primary Angle Closure Suspects: A Swept Source Anterior Segment Optical Coherence Tomography Study. J Glaucoma. 2020 Jul;29(7):521-528. doi: 10.1097/IJG.0000000000001506. PMID 32224802